CLINICAL TRIAL: NCT02461420
Title: Mapping the Genotype, Phenotype, and Natural History of Phelan-McDermid Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Phelan-McDermid Syndrome Foundation (Other)
Responsible Party: Principal Investigator, Mustafa Sahin, Professor of Neurology, Harvard Medical School, Boston Children's Hospital
Other Study IDs: P00013300; 1U54NS092090 (NIH)
Record Dates: First submitted 2015-05-11; First posted 2015-06-03 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Phelan-McDermid Syndrome; Autism Spectrum Disorder; Intellectual Disability
Keywords: Phelan-McDermid Syndrome; PMS; Genotype; Phenotype; Natural History; Mapping; 22q13 Deletion Syndrome; SHANK3; Autism Spectrum Disorder; ASD; Intellectual Disability; ID; EEG
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome; Autism Spectrum Disorder; Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw for future correlative studies in the PMS Biorepository of the Developmental Synaptopathies Consortium
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Phelan-McDermid Syndrome: Phelan-McDermid Syndrome

SUMMARY:
The purpose of this study is to comprehensively characterize PMS using standardized medical, cognitive, and behavioral measures and to track the natural history of the syndrome using repeated longitudinal assessments. In addition, this study will be aiming to identify biomarkers using neuroimaging, including diffusion tensor imaging and identify genetic factors which contribute to diverse phenotypes in patients with PMS.

DETAILED DESCRIPTION:
Phelan-McDermid syndrome (PMS) or 22q13 Deletion syndrome, caused by a loss of one copy of the SHANK3 gene, is characterized by global developmental delay/intellectual disability, motor skills deficits, delayed or absent speech, and autism spectrum disorder. The goal of this study is to understand more about the PMS phenotype and the biological pathways associated with ID and ASD in the disorder, and to establish the foundation for future clinical trials in PMS and in other ID/ASD-associated disorders that share signaling pathways with PMS.

Individuals with PMS will be asked to participate in this study if they are 18 months or older with pathogenic deletions or mutations of the SHANK3 gene at time of enrollment, as well as healthy controls. Both males and females will be asked to participate. Additionally, to be eligible for study participation, individuals' primary communicative language must be English. Parents and unaffected siblings may also be asked to consent to have blood drawn for analysis.

The study involves 3 on site visits over 2 years. Study visits involve a physical exam, medical history questions, blood work and neuropsychological assessments. A subset of participants between the ages of 2 and 11 years old will take part in the EEG portion of the study. Individuals who have a clinically indicated MRI will have an option to provide routine clinical scans for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals older than 18 months of age with pathogenic deletions or mutations of the SHANK3 gene
* English speaking individuals

Exclusion Criteria:

* Has taken an investigational drug as part of another research study, within 30 days prior to study enrollment
* For subjects involved in imaging biomarker assessment: contraindications to 3T MRI scanning, such as metal implants/non-compatible medical devices or medical conditions, including vagus nerve stimulator
* For subjects involved in EEG/ ERP biomarker assessment: contraindications to EEG/ERP, such as uncooperative or destructive behaviors preventing lead placement or capture by ERP/VEP equipment. Under age 2 or over age 11 at the time of enrollment.
* Unwilling or unable to comply with study procedures and assessments

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 190 subjects with PMS will be enrolled across the 6 sites for this study
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2015-05; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive ability at 12 months | 12 months
  Using Mullen Scales for Early Learning or Stanford Binet-5 to measure global cognitive ability
Change in adaptive behavior at 12 months | 12 months
  Using Vineland Adaptive Behavior Scales to measure adaptive behavior
Change in language abilities at 12 months | 12 months
  Using composite of Mullen Subscales, Vineland Subscales and Macarthur Bates Communication Developmental Inventory to measure language
Change in motor functioning at 12 months | 12 months
  Using composite of Mullen Subscales and Vineland Subscales to measure motor functioning
Change in autism symptoms at 12 months | 12 months
  Using composite of Autism Diagnostic Observation Schedule and Repetitive Behavior Scales-Revised to measure autism
Change in global cognitive ability at 24 months | 24 months
  Using Mullen Scales for Early Learning or Stanford Binet-5 to measure global cognitive ability
Change in adaptive behavior at 24 months | 24 months
  Using Vineland Adaptive Behavior Scales to measure adaptive behavior
Change is language abilities at 24 months | 24 months
  Using composite of Mullen Subscales, Vineland Subscales and Macarthur Bates Communication Developmental Inventory to measure language
Change in motor functioning at 24 months | 24 months
  Using composite of Mullen Subscales and Vineland Subscales to measure motor functioning
Change in autism symptoms at 24 months | 24 months
  Using composite of Autism Diagnostic Observation Schedule and Repetitive Behavior Scales-Revised to measure autism

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kolevzon, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - National Institutes of Health, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Derived] Bassell J, Srivastava S, Prohl AK, Scherrer B, Kapur K, Filip-Dhima R, Berry-Kravis E, Soorya L, Thurm A, Powell CM, Bernstein JA, Buxbaum JD, Kolevzon A, Warfield SK, Sahin M; Developmental Synaptopathies Consortium. Diffusion Tensor Imaging Abnormalities in the Uncinate Fasciculus and Inferior Longitudinal Fasciculus in Phelan-McDermid Syndrome. Pediatr Neurol. 2020 May;106:24-31. doi: 10.1016/j.pediatrneurol.2020.01.006. Epub 2020 Jan 31. PMID 32107139
- [Derived] Srivastava S, Scherrer B, Prohl AK, Filip-Dhima R, Kapur K, Kolevzon A, Buxbaum JD, Berry-Kravis E, Soorya L, Thurm A, Powell CM, Bernstein JA, Warfield SK, Sahin M; Developmental Synaptopathies Consortium. Volumetric Analysis of the Basal Ganglia and Cerebellar Structures in Patients with Phelan-McDermid Syndrome. Pediatr Neurol. 2019 Jan;90:37-43. doi: 10.1016/j.pediatrneurol.2018.09.008. Epub 2018 Sep 21. PMID 30396833